CLINICAL TRIAL: NCT06459661
Title: The Bowel Movement Monitoring (BoMoMo) Study: An Exploration of the Relationship Between Intake of Unrefined, Intact Plant Foods and Faecal Output
Brief Title: The Bowel Movement Monitoring (BoMoMo) Study
Acronym: BoMoMo
Status: Recruiting | Type: Observational
Sponsor: Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Beverley O'Hara, Lecturer (Nutrition), Leeds Beckett University
Other Study IDs: BO01
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Dietary Exposure
MeSH Terms: interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diet — Intake of unrefined, intact plant foods

SUMMARY:
The link between what people eat and how it affects faecal output (poo) has been understudied. Most of the research that has looked at the link between diet, bowel movements and overall health has studied different types of fibre extracted from foods (e.g., fibre extracted from carrots), rather than foods in the form that they are consumed.

It is necessary for scientists to investigate the relationship between food as people usual eat it (e.g., a carrot) and bowel movements, as this information is key to understanding the relationship between what people eat and overall health.

The investigators would like to understand the relationship between intake of certain foods and faecal output. This will help to develop a chart, similar to the United Kingdom National Health Service urine colour hydration chart. The chart will allow people to know, by looking at their poo, whether they are eating enough of the foods that will keep them healthy. By monitoring and measuring participants' bowel movements, and providing information about diet, participants will provide the data we need for this research.

DETAILED DESCRIPTION:
Participants will complete a 5-day estimated food record and weigh, characterise and photograph each stool for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years.
* Healthy as determined from self-reported medical history or when no relevant medical condition exists.
* Stool frequency of 3 to 21 times per week.
* Able to attend a session in person at City Campus or Headingley Campus, Leeds Beckett University, or City Campus, Sheffield Hallam University.
* For women: Use of contraceptive methods or not planning to become pregnant for the duration of the study.
* Able to understand and be willing to sign the informed consent form, and to follow all the study procedures and requirements.

Exclusion Criteria:

* Food allergy or intolerance
* Currently dieting to lose weight
* For women: Pregnancy, lactation
* Bowel disease
* Use of medicine causing constipation
* Abnormal gastro-intestinal (gut) function or structure such as malformation, angiodysplasia or active peptic ulcer
* History of gastro-intestinal surgery with permanent effect (e.g., surgical treatment of obesity)
* Active inflammatory bowel disease, coeliac disease, chronic pancreatitis, or other disorder potentially causing malabsorption
* Currently experiencing or been diagnosed with gastro-intestinal symptoms (e.g., abdominal pain/cramps, heartburn, stomach acid/reflux, nausea, vomiting, abdominal rumbling, bloating, belching, excess gas/wind)
* Active constipation (i.e., currently constipated).
* Active Irritable Bowel Syndrome
* Currently experiencing disordered eating
* Current use of laxatives
* Current use or within the previous 3 months use of prescription or over-the-counter medication that has the potential of affecting gut bacteria including food supplements (specific medications will be assessed on an individual basis).
* Use of antibiotics or pain medication containing opiates or morphine currently or within the previous 3 months.
* Use of opioid drugs of abuse (e.g., heroin, fentanyl) currently or within the previous 3 months.
* Consumption of more than 21 units of alcohol per week (men)/ more than 14 unit of alcohol per week (women).
* Malignancy/cancer which is currently active or in remission for less than 2 years after treatment.
* Currently experiencing a psychiatric disorder or a condition related with your mental health that impacts on your daily life (e.g., major depression, bipolar disorders).
* Currently engaging in intense physical activity more than 3 times per week (assessed on an individual basis).
* Presenting a psychological or linguistic incapability to sign the informed consent/ Investigator considers the subject unlikely to comply with study procedures, restrictions, and requirements.
* Parallel participation in another research project which involves dietary intervention/other clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Faecal weight | 5 days
  Average weight of faeces

SECONDARY OUTCOMES:
Faecal bulk | 5 Days
  Volume of faeces

OTHER OUTCOMES:
Time to pass stool | 5 Days
  Number of seconds taken to pass stool
Stool type | 5 Days
  Average Bristol Stool Form Scale type (Type 1-7 nominal scale; types 3,4,5 are considered the 'normal range')

CONTACTS AND LOCATIONS:
Locations (1):
- Beverley O'Hara, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided